CLINICAL TRIAL: NCT01104909
Title: Randomized Clinical Trial Evaluating Different Protocols for Improving the Way of Getting the Best Dry Weight for Hemodialysis Patients, Looking for Blood Pressure Control, Measured by ABPM
Brief Title: How to Get a Better Dry Weight in End-stage Renal Disease (ESRD) Population for Improving Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade de Passo Fundo (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Darlan Martins Lara, Universidade Federal do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DryWeightESRDxBloodPressure; ESRD; Blood Pressure; Dry weight
Record Dates: First submitted 2010-04-13; First posted 2010-04-16 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Blood Pressure; End Stage Renal Disease; Hemodialysis
Keywords: Dry weight; Blood Pressure; Chronic Kidney disease
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinical dry weight (Active Comparator): Group which the dry weight will be assessed based on clinical examination.
  Interventions: Procedure: Clinical
- Bioimpedance (Active Comparator): Group which the dry weight will be assessed by bioimpedance data.
  Interventions: Device: electrical bioimpedance

INTERVENTIONS:
Procedure: Clinical — Each patient will be submitted a clinical evaluation, considering signals of overload.
  Arms: Clinical dry weight
Device: electrical bioimpedance — From electrical bioimpedance data, will be fixed a revised dry weight for each patient.
  Arms: Bioimpedance

SUMMARY:
End-stage renal disease (ESRD) is a common clinical condition. In this population, the prevalence of systemic hypertension is high and its adequate control can determinate the outcome.

The first step for a good control of blood pressure in renal patients is adjusting his/her dry weight. Actually, dry weight is assessed based on clinical examination and blood pressure.

The electrical bioimpedance is a simple and portable device. The investigators design a randomized clinical trial for evaluating two ways of getting the best dry weight for hemodialysis patients.

A basal 24h ABPM will be taken before the randomization. Then, 2 weeks later the dry weight be revised, the investigators will get a second 24h ABPM.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) is a common clinical condition over the world. In this population, the prevalence of systemic hypertension is high and its adequate control can determinate the outcome.

The first step for a good control of blood pressure is giving a dry weight for the patient. We can understand dry weight or target weight as that one which the patient feels comfortable and there aren't clinical signals of volemic overload as edema, dyspnea, orthopnea, jugular turgency, hepatomegalia. Classically, the dry weight is assessed based on clinical examination, blood pressure and experience of hemodialysis staff.

The electrical bioimpedance is a very simple method that possibilities access the corporal compartments, including the body water, using a small and not expensive portable device.

Trying to study new forms for getting the ideal dry weight, we design a randomized clinical trial for evaluating two ways of getting a dry weight for hemodialysis patients.

One group will be dry weight fixed by bioimpedance data and in another group the dry weight will by a clinical protocol.

We will take a 24h ABPM basal from all patients before the randomization. Then, 2 weeks later the dry weight be revised, a second ABPM will be taken. The results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD, clinically stable, under hemodialysis therapy at two clinics in the North of Rio Grande do Sul.

Exclusion Criteria:

* Clinical unstability, like: infection in course ou recent acute cardiovascular disease (less then 3 months).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-05 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Diastolic and systolic blood pressure assessed by ABPM | after 2 weeks
  A basal measure will be taken at the start point. Then, the dry weight will be evaluated by clinical or BIA method. After 2 weeks of tree times-week sections of hemodialysis under the revised dry weight, a second measure of ABPM will be performed.

SECONDARY OUTCOMES:
intradialytic signals and/or symptoms | during two weeks
  the intradialytic signals and/or symptoms will be assessed by dialysis registers, before and after de revision of dry weight

CONTACTS AND LOCATIONS:
Overall Officials: Darlan M Lara, MD MsC, Principal Investigator — Fedral University of Rio Grande do Sul; Miguel Gus, MD PhD., Study Chair — Federal University of Rio Grande do Sul
Locations (1):
- Darlan Martins Lara, Carazinho, Rio Grande do Sul, Brazil